CLINICAL TRIAL: NCT01394848
Title: EndothelIal progeNitor Cell Capture steNt With 1-mOnth Dual Antiplatelet Therapy Versus eVerolimus-eluting Stent With stAndard 12-month Dual anTIplatelet Therapy in Elderly (≥ 70 Year) With Stable corONary Artery Disease - INNOVATION Trial
Brief Title: Safety and Efficacy Study of Endothelial Progenitor Cell Capture Stent With 1 Months Dual Antiplatelet Therapy
Acronym: INNOVATION
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Previous other study including EPC capture stent raised the issue of safety (significant high incidence of instent restenosis)
Sponsor: Yonsei University (Other)
Collaborators: OrbusNeich (Industry); Yuhan Corporation (Industry)
Responsible Party: Principal Investigator, Seung-Hwan Lee, Professor, Yonsei University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: INNOVATION_v5.0
Record Dates: First submitted 2011-07-11; First posted 2011-07-14 (Estimated); Last update posted 2013-12-04 (Estimated); Status verified 2013-12

CONDITIONS: Stable Angina
MeSH Terms: conditions — Angina, Stable | interventions — Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Genous stent group (Active Comparator): Genous stent (Endothelial progenitor cell capture stent) insertion in elderly patients with stable coronary artery disease
  Interventions: Device: Endothelial cell capture stent with 1 month clopidogrel
- Xience stent group (Active Comparator): Xience Prime V stent (everolimus eluting stent) insertion in elderly patients with stable coronary artery disease
  Interventions: Device: Everolimus eluting stent with 12 month clopidogrel
- Atorvastatin 20mg group (Active Comparator)
  Interventions: Drug: Atorvastatin 20mg loading
- Atorvastatin 80mg group (Active Comparator)
  Interventions: Drug: Atorvastatin 80mg loading

INTERVENTIONS:
Device: Endothelial cell capture stent with 1 month clopidogrel — 75mg PO clopidogrel per day for 1 months
  Other Names: Genous stent
  Arms: Genous stent group
Device: Everolimus eluting stent with 12 month clopidogrel — 75mg PO clopidogrel per day for over 12 months
  Other Names: Xience stent
  Arms: Xience stent group
Drug: Atorvastatin 20mg loading — Atorvastatin 20mg loading before index percutaneous coronary intervention
  Other Names: Atorvastatin
  Arms: Atorvastatin 20mg group
Drug: Atorvastatin 80mg loading — Atorvastatin 80mg loading before index percutaneous coronary intervention
  Other Names: Atorvastatin
  Arms: Atorvastatin 80mg group

SUMMARY:
Thanks to rapid reendothelialization derived from the pro-healing property of the EPC capture stent, 1-month dual antiplatelet therapy (DAPT) is recommended after EPC capture stent implantation. Shorter maintenance of dual antiplatelet therapy might minimize the risk for stent thrombosis in cases of discontinuation of antiplatelet regimen and prevent wasteful medications and bleeding complications related with dual antiplatelet therapy. Thus, the EPC capture stent might be valuable for the elderly because they are vulnerable to premature discontinuation of DAPT.

On the other hand, statin upstream therapy has gained popularity because it seems to reduce periprocedural myocardial injury especially in ACS through its pleiotrophic effect like plaque stabilization. However, the benefit of pretreatment of statin in patients with stable angina remains controversial. It is reported that statin administration could increase EPC level by accelerated differentiation towards the endothelial progenitor lineage.

We hypothesize that the EPC capture stent with 1-month dual antiplatelet therapy is non-inferior to DES in the elderly subjects with stable coronary artery disease. To test this hypothesis, we will perform a multi-center, randomized, prospective trial aimed at demonstrating the efficacy and safety of the EPC capture stent with 1-month DATP versus EES with standard 12-month DAPT in elderly patients with stable coronary occlusive disease in real world practice.

DETAILED DESCRIPTION:
Drug-eluting stents (DES) have improved angiographic and clinical outcomes in patients with the complex coronary lesions and high risks by markedly reducing the neointimal hyperplasia following stent implantation in comparison to bare-metal stents (BMS). Although the concerns about long-term safety and the occurrence of stent thrombosis following DES implantation had been raised, the recent DES-registry studies have reported that DES did not increase the risk of death or stent thrombosis during follow-up, as compared with BMS. However, currently, the fatal events related with stent thrombosis still occur and are the major limitation of the use of DES. Especially, late or very late thrombosis after DES implantation is an uncommon but life-threatening fatal complication presented with sudden death or myocardial infarction (MI).

The most powerful predictor for stent thrombosis is the discontinuation of clopidogrel. Then, under these circumstances, the prolonged dual antiplatelet therapy is now recommended, irrespective of each precise consideration according to the types of DES, lesion complexity, or clinical characteristics. Although the prolonged antiplatelet therapy can prevent stent thrombosis, it might cause other problems such as combined bleeding complications, high cost due to prolonged use, and unnecessary maintenance of medication. The stratified strategies regarding antiplatelet therapy according to the lesion complexity or high risks such as diabetes or acute coronary syndrome, which were regarded as the most prominent predictors for stent thrombosis, should be required. Another difficult problem of DES in real world practice is how we can manage the cases in which clopidogrel should be discontinued due to unexpected minor and major operations or invasive procedures. Because there have been no available substitutes as a bridging therapy of clopidogrel until operation, many advisory groups recommend to hold on off elective non-cardiac surgery 12 months after DES implantation. If not, BMS implantation is strongly recommended for patients with high risk of bleeding or scheduled unavoidable surgery within the next 12 months. Especially in the elderly, premature discontinuation of DAPT within 12 months after PCI may occur due to combined co-morbid disease requiring surgical intervention, decreased drug compliance, or occurrence of gastrointestinal bleeding.

Recently, many attempts to elucidate the mechanism of stent thrombosis have been performed. Finn AV et al. have reported from the human autopsies of DES that the most powerful histological predictor of stent thrombosis was endothelial coverage and suggested stent strut coverage as a marker of endothelialization. After then, the more concerns have been focused on the healthy healing after DES implantation, in spite of relatively higher late lumen loss. As a result, when antiplatelet therapy should be discontinued, DES with a healthy healing might be more preferred, instead of efficient DES with a lower late lumen loss.

In the view of these points, in spite of actual higher late lumen loss, Endothelial Progenitor Cell (EPC) Capture Stent (GENOUS™ Bio-engineered R stent™, OrbusNeich) could be more beneficial and safer than DES because of its low risk for stent thrombosis due to more rapid endothelialization and its resulting short-term use of dual antiplatelet. EPC capture stent has antibodies immobilized on the stent surface to capture circulating endothelial progenitor cells leading to accelerated natural healing. Theoretically, the EPC capture stent has two benefits. It establish functional endothelium, therefore no longer term anti-platelet therapy is required. Second, EPC capture stent may minimizes restenosis, because it establishes healthy endothelium which expresses vasoactive compounds, such as nitric oxide, which modulates neo-intimal hyperplasia and thus restenosis.

Thanks to rapid reendothelialization derived from the pro-healing property of the EPC capture stent, 1-month dual antiplatelet therapy (DAPT) is recommended after EPC capture stent implantation. Shorter maintenance of dual antiplatelet therapy might minimize the risk for stent thrombosis in cases of discontinuation of antiplatelet regimen and prevent wasteful medications and bleeding complications related with dual antiplatelet therapy. Thus, the EPC capture stent might be valuable for the elderly because they are vulnerable to premature discontinuation of DAPT.

On the other hand, statin upstream therapy has gained popularity because it seems to reduce periprocedural myocardial injury especially in ACS through its pleiotrophic effect like plaque stabilization. However, the benefit of pretreatment of statin in patients with stable angina remains controversial. It is reported that statin administration could increase EPC level by accelerated differentiation towards the endothelial progenitor lineage.

We hypothesize that the EPC capture stent with 1-month dual antiplatelet therapy is non-inferior to DES in the elderly subjects with stable coronary artery disease. To test this hypothesis, we will perform a multi-center, randomized, prospective trial aimed at demonstrating the efficacy and safety of the EPC capture stent with 1-month DATP versus EES with standard 12-month DAPT in elderly patients with stable coronary occlusive disease in real world practice.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥70 years patients with coronary artery disease (≤stable angina CCS III, Unstable angina IIb
* patients with signed informed consent
* significant coronary artery stenosis (>50%) considered for coronary stenting
* Reference vessel diameter of 2.5 to 4.0 mm

Exclusion Criteria:

* The patient has a known hypersensitivity or contraindication to any of the following medications: Heparin, Aspirin, Clopidogrel, Everolimus, Contrast media (Patients with documented sensitivity to contrast media which can be effectively premedicated with steroids and diphenhydramine [e.g. rash] may be enrolled. Those with true anaphylaxis to prior contrast media, however, should not be enrolled.)
* Systemic (intravenous) Everolimus use within 12 months
* The patients who are receiving anticoagulants or anti-platelet medications besides aspirin & clopidogrel
* History of bleeding diathesis or known coagulopathy (including heparin-induced thrombocytopenia), or refuses blood transfusions
* Baseline hemogram with Hb<10g/dL or PLT count <100,000/μL
* Severe Hepatic dysfunction (≥ 3 times normal reference values)
* Significant renal dysfunction (Serum creatinine ≥ 2.0 mg/dl)
* Gastrointestinal or genitourinary bleeding within the prior 3 months, or major surgery within 2 months
* Patients with LV systolic dysfunction (LVEF<40%) or in cardiogenic shock
* Non-cardiac co-morbid conditions are present with life expectancy <1 year or that may result in protocol non-compliance (per site investigator's medical judgment)
* Patients who are actively participating in another drug or device investigational study, which have not completed the primary endpoint follow-up period
* An elective surgical procedure is planned that would necessitate interruption of DAPT during the first 12 months post enrollment

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 1 (Actual)
Dates: Start 2011-10; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Major adverse cardiovascular events | 12 months
  The incidence of the composite of cardiovascular death, non-fatal myocardial infarction (MI), target lesion revascularization (TLR), or stent thrombosis following randomly assigned coronary stent implantation

SECONDARY OUTCOMES:
Each component of the primary composite endpoint at 12 months | 12 months
In-stent late loss and angiographic pattern of restenosis at 13 months | 13 months
In-sent and in-segment % diameter stenosis (%DS) at 13 months | 13 months
Overall incidence of deferring or declining the request to discontinue dual antiplatelet between 1-12 months due to major and minor operations or invasive procedures | 12 months
Cost-reducing effect according the duration of duration of anti-platelet therapy | 12 months
Periprocedural myocardial infarction | 12 months
Bleeding defined by Bleeding Academic Research Consortium (BARC) | 12 months
  Bleeding Academic Research Consortium Definition for Bleeding Type 0 to Type 5

CONTACTS AND LOCATIONS:
Overall Officials: Seung-Hwan Lee, MD, PhD, Principal Investigator — Yonsi university Wonju college of medicine, Wonju christian hospital
Locations (1):
- Yonsei university Wonju College of Medicine, Wŏnju, Gangwon-do, South Korea